CLINICAL TRIAL: NCT03265587
Title: FARCE Study: Feng Shui And Emotional Response in the Critical Care Environment
Brief Title: Feng Shui And Emotional Response in the Critical Care Environment Study
Acronym: FARCE
Status: Completed | Type: Observational
Sponsor: Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16/HRA/5855
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Feng Shui
Keywords: Feng Shui; Inner harmony; Chi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Orientation 1: Nursing staff allocated to a bed space with orientation 1
  Interventions: Other: No intervention
- Orientation 2: Nursing staff allocated to a bed space with orientation 2
  Interventions: Other: No intervention
- Floater / Control group: Nursing staff not allocated to a bed space with an orientation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Objective: To assess whether the feng shui of critical care bed spaces affects the inner harmony of nursing staff Design: Prospective cohort study Setting: Doncaster critical care department Participants: Critical care nursing staff Main outcome measures: To assess self-reported chi scores and their response to feng shui, cake ingestion and ghost sightings

DETAILED DESCRIPTION:
Feng Shui Feng shui is an ancient Chinese system that governs the arrangement and orientation of objects in a room, in relation to the flow of energy called chi or qi. The flow of chi in a room or building may have beneficial or undesirable effects on a persons' feelings and inner harmony. Each feeling is associated with an element: fire, water, wood, earth and metal. These elements are used to describe the colours and shapes in the surroundings. For example fire could be represented as a candle for many reasons; the flame, warmth generated from the flame and red colour.

Bagua A bagua is a tool used to map an area to facilitate the flow of chi. A traditional bagua is octagonal, each of the eight segments associated with a feeling and therefore an element, shape and colour. The traditional bagua is aligned to the compass before an area is mapped out.The western bagua uses a nine panelled grid, with each panel associated with a feeling and therefore an element, shape and colour.The base of the grid is aligned against the wall of a room which has the main entrance contained within it. The room can then be divided into nine sections, each corresponding to a bagua panel. Objects that possess qualities of an element can then be rearranged to promote the flow of chi in a certain area of a room.

Nurturing and destructive relationships There are nurturing and destructive relationships between the elements, that affect the flow of chi and therefore the feelings of the affected element.For example an earth object placed in an area associated with metal will increase the flow of chi in this area and increase the feelings associated with it. Equally if a fire object is placed in an area associated with metal, there will be a negative impact on the flow of chi and therefore the a reduction in the feelings in this area. Using the above principles of feng shui it is possible to re-arrange a room to enhance the flow chi and achieve positive influence for ones feelings. It may not be possible to completely re-arrange a room due to fixed structures such as a window, radiator etc. In this case a bagua and knowledge of the nurturing and destructive cycles can be used to make adjustments to get the best possible flow of chi.

Critical care Critical care departments can be intensive places to work. In addition to the usual hospital equipment such as a bed, locker and table, critical care bed spaces have several extra pieces of equipment including a ventilator and stacks for infusion pumps. By mapping and scoring bed space orientations, we hypothesized that it is possible to predict how nursing staff should feel working in these bed spaces. The purpose of this study was to determine whether the principles of feng shui apply to critical care bed spaces and therefore affect the inner harmony of nursing staff during a shift.

The critical care department to be studied contains 20 beds that are used for a mix of level two or three care depending upon patient need and nursing staff capacity. Of these beds, 15 are split almost equally into two orientations. A plan of each orientation will be divided into nine sections to correspond to a bagua panel. Each item of equipment will be assigned a feng shui element based upon its shape or colour. Using a bagua, the feng shui of each bed space will be mapped. For each bagua panel a +1 will be awarded for each piece of equipment that positively influenced chi either directly or indirectly through the nurturing cycle. Conversely a -1 will be awarded for each piece of equipment that negatively influenced chi either directly or indirectly through the destructive cycle. The points awarded in each panel will then be added together to give a feng shui score for that panel. The feng shui score will be limited to -5 and +5. This score will then be converted to a 0-10 'chi score' for nurse self-assessment and to allow data analysis.

For the purpose of our study we assume that a positive score would result in a positive flow of chi and therefore positively affect the feeling or attribute associated with that panel for a nurse working at that bed space. We assume the opposite would be true of a negative score.

Critical care nursing staff will be allocated to bed spaces by the nursing coordinator, the allocation may be based upon nursing skill mix. Nursing staff will be asked to voluntarily complete a questionnaire towards the end of their shift.

Data Questionnaires will be distributed to all participants. The questionnaire requires participants to self-assess their chi by rating nine feelings associated with the bagua and their overall inner harmony from 0 to 10 (Table 1). Participants will be blinded to the feng shui scoring of their bed space. Nursing staff who are not assigned to a bed space will also be asked to fill in the questionnaire to act as a control group.

The investigators have previously observed that cake has a positive effect on nursing staff mood. The study hospital is also well known for ghost sightings which may result in negative mood. Therefore the questionnaire also asks if the nursing staff have encountered either of these potentially confounding factors. Questionnaires will collected and stored until after the study period expired.

There will be no patient participation Statistical analysis will be performed using IBM SPSS (version 22). A p-value of <0.05 was regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Critical care nursing staff volunteering for the study

Exclusion Criteria:

* Refusal to participate
* Critical care nursing staff assigned to non-study bed spaces
* Critical care nursing staff assigned to more than one bed spaces orientation per shift

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Doncaster Royal Infirmary critical care nursing staff and health care assisants
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
To measure the effects of feng shui on critical nursing staff inner harmony | Nursing shifts last 12 hours - questionnaires will be voluntarily completed at the end of a shift. The trial will run over a 14 day period.
  Each bed space orientation has a calculated bed space feng shui score. This will be used to predict how nursing staff feel at the end of their shift. Nursing staff will be given a questionnaire to voluntarily fill in asking them to rate 10 feelings. Nursing staff will have the option of rating each feeling from 0 to 10. The resulting nurse self assessment score will then be compared to the calculated bed space feng shui score.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Charles, Study Director — National Health Service, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Definition of feng shui — http://www.dictionary.com/browse/feng-shui
- See also: Information regarding feng shui — https://en.wikipedia.org/wiki/Feng_shui
- See also: Information regarding feng shui — http://fengshuiforreallife.com